CLINICAL TRIAL: NCT01805492
Title: Global Profiling of Gene and Protein Expression Associated With Coronary Heart Disease Reversal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Windber Research Institute (Other)
Responsible Party: Principal Investigator, Darrell L Ellsworth, Senior Director, Integrative Cardiac Health Program, Windber Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRI-03-03; MDA W81XWH-05-2-0075 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2013-02-21; First posted 2013-03-06 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Heart Diseases; Cardiovascular Diseases
Keywords: Heart diseases; Cardiovascular diseases; Lifestyle modification; Diet; Exercise
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Dr. Dean Ornish Program for Reversing Heart Disease
  Interventions: Behavioral: Dr. Dean Ornish Program for Reversing Heart Disease
- Control (No Intervention): Non-intervention controls retrospectively matched to intervention participants

INTERVENTIONS:
Behavioral: Dr. Dean Ornish Program for Reversing Heart Disease — Prospective, nonrandomized clinical intervention to stabilize or reverse progression of heart disease through changes in lifestyle. Lifestyle intervention consisted of four components: 1) a very low fat vegetarian diet (<10% of calories from fat); 2) 180 minutes/week of moderate aerobic exercise; 3) one hour of stress management each day; and 4) weekly group support sessions.
  Arms: Intervention

SUMMARY:
The purpose of this study is to characterize changes in gene and protein expression in peripheral blood in patients with, or at risk for, heart disease during an intensive lifestyle modification program.

DETAILED DESCRIPTION:
This project will use an integrated approach that examines DNA variation and the functional products of genes at both the messenger RNA (mRNA) and protein levels to provide a global view of molecular changes associated with drastic lifestyle modifications designed to reverse coronary heart disease (CHD). DNA variants and/or changes in gene and protein expression associated with CHD reversal may provide important clues to understanding molecular mechanisms of subclinical CHD development and progression.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of coronary artery disease (CAD)
* stable angina
* angioplasty
* evidence of >50% luminal narrowing on coronary angiogram
* acute myocardial infarction
* bypass surgery
* stent placement OR
* two or more CAD risk factors
* systolic pressure >140 mm Hg or diastolic pressure >90 mm Hg)
* high total cholesterol (>200 mg/dL)
* physician diagnosed diabetes
* body mass index (BMI) >30
* family history of heart disease in parents or siblings
* 21 years of age or older
* mentally competent to provide informed consent

Exclusion Criteria:

* known history of autoimmune disease
* systemic/chronic disease requiring chemotherapy or long term treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2000-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Change in body mass index | Baseline, 12 weeks, 52 weeks
  Change in BMI from baseline to 12 weeks and from baseline to 52 weeks

SECONDARY OUTCOMES:
Change in blood pressure | Baseline, 12 weeks, 52 weeks
  Change in BP from baseline to 12 weeks and from baseline to 52 weeks
Change in lipids | Baseline, 12 weeks, 52 weeks
  Change in HDL-, LDL-, total cholesterol, and triglycerides from baseline to 12 weeks and from baseline to 52 weeks
Change in exercise capacity | Baseline, 12 weeks, 52 weeks
  Change in exercise capacity from baseline to 12 weeks and from baseline to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Darrell L Ellsworth, PhD, Principal Investigator — Windber Research Institute
Locations (1):
- Windber Medical Center, Windber, Pennsylvania, United States

REFERENCES:
- [Result] Ellsworth DL, O'Dowd SC, Salami B, Hochberg A, Vernalis MN, Marshall D, Morris JA, Somiari RI. Intensive lifestyle modification: impact on cardiovascular disease risk factors in subjects with and without clinical cardiovascular disease. Prev Cardiol. 2004 Fall;7(4):168-75. doi: 10.1111/j.1520-037x.2004.3332.x. PMID 15539963
- [Result] Vizza J, Neatrour DM, Felton PM, Ellsworth DL. Improvement in psychosocial functioning during an intensive cardiovascular lifestyle modification program. J Cardiopulm Rehabil Prev. 2007 Nov-Dec;27(6):376-83; quiz 384-5. doi: 10.1097/01.HCR.0000300264.07764.84. PMID 18197071
- [Result] Decewicz DJ, Neatrour DM, Burke A, Haberkorn MJ, Patney HL, Vernalis MN, Ellsworth DL. Effects of cardiovascular lifestyle change on lipoprotein subclass profiles defined by nuclear magnetic resonance spectroscopy. Lipids Health Dis. 2009 Jun 29;8:26. doi: 10.1186/1476-511X-8-26. PMID 19563671
- [Result] Voeghtly LM, Neatrour DM, Decewicz DJ, Burke A, Haberkorn MJ, Lechak F, Patney HL, Vernalis MN, Ellsworth DL. Cardiometabolic risk reduction in an intensive cardiovascular health program. Nutr Metab Cardiovasc Dis. 2013 Jul;23(7):662-9. doi: 10.1016/j.numecd.2012.01.012. Epub 2012 May 26. PMID 22633795
- [Derived] Ellsworth DL, Croft DT Jr, Weyandt J, Sturtz LA, Blackburn HL, Burke A, Haberkorn MJ, McDyer FA, Jellema GL, van Laar R, Mamula KA, Chen Y, Vernalis MN. Intensive cardiovascular risk reduction induces sustainable changes in expression of genes and pathways important to vascular function. Circ Cardiovasc Genet. 2014 Apr;7(2):151-60. doi: 10.1161/CIRCGENETICS.113.000121. Epub 2014 Feb 21. PMID 24563419
- See also: Windber Research Institute home page — http://www.wriwindber.org/